CLINICAL TRIAL: NCT06673355
Title: Comparative Study of Different Supra-structure Materials in Digitally Designed Full-arch Implant-supported Prosthesis. (Bone Changes and Teeth Wear Analysis) - a Randomized Clinical Trial
Brief Title: "Comparative Study of Supra-Structure Materials in Full-Arch Implant Prosthetics: a Randomized Clinical Trial"
Acronym: CSDSMDA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, HEBA ELSARRIF, Principal Investigator - Lecturer of Removable Prosthodontics, Misr University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RECO6U/2024
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Edentulous Mandible
Keywords: all on 4 full arch restorations in the mandible

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patients will receive frameworks made of high-performance polymer (Experimental): patients will receive frameworks made of high-performance polymer filled with nano zirconia and carbon, the framework will be digitally produced by the milling technology using a dental CNC machine. the bone changes and occlusal wear will be assessed at the time of insertion (as a baseline), after 6 months and after 12 months.
  Interventions: Other: dental implant prosthesis
- patients will receive frameworks made of porcelain fused to titanium (Active Comparator): patients will receive frameworks made of porcelain fused to titanium, the titanium will be produced digitally by 3d printing using the selective laser melting technology. Bone changes and wear of occlusal surfaces will be assessed at time of insertion (baseline, after 6 months and after 12 months
  Interventions: Other: dental implant prosthesis

INTERVENTIONS:
Other: dental implant prosthesis — patients will receive frameworks made of high-performance polymer filled with nano zirconia and carbon

SUMMARY:
after the implants' osseointegration period (4 months), digital scans will be taken for the implant positions and the STL files will be stored and sent for the CAD software to design a full arch restoration. Two types will be constructed, Group I patients will receive porcelain fused to titanium frameworks, and Group II will receive a framework made of high-performance polymer filled with nano-zirconia and carbon. After the installation of the frameworks, the bone height changes and the wear of the occlusal surfaces will be monitored at baseline, after 6 months and 12 months post insertion.

DETAILED DESCRIPTION:
After the implants' osseointegration period of four months, a series of steps will be undertaken to ensure the precise design and implementation of the full-arch restorations.

First, digital scans of the implant positions will be conducted using advanced scanning technology. These scans will accurately capture the spatial orientation and positioning of the implants within the jaw. The resulting STL (Standard Tessellation Language) files, which represent the 3D geometry of the scanned implants, will be securely stored and transmitted to computer-aided design (CAD) software. This software will facilitate the design process for the full-arch restorations.

In this study, two distinct types of full-arch frameworks will be constructed for the participants, who will be divided into two groups based on the material used.

* **Group I** will receive frameworks made of porcelain fused to titanium (P/FtTi). This material is known for its strength, durability, and aesthetic qualities, providing a reliable option for prosthetic restorations.
* **Group II** will receive frameworks crafted from a high-performance polymer enhanced with nano-zirconia and carbon fillers. This innovative material is designed to offer superior mechanical properties, including increased strength and reduced wear while being lightweight and biocompatible.

Once the frameworks are installed in the patient's mouth, the study will focus on monitoring the changes in bone height and the wear of the occlusal surfaces over time. Measurements will be taken at three key intervals: baseline ( time of framework fixation), and then again at six months and twelve months post-insertion.

This monitoring will involve radiographic assessments using CBCT and clinical evaluations to quantify any bone resorption around the implants and to assess the wear patterns of the occlusal surfaces using the intraoral scanner, the STL files of the scans will be superimposed on a software (Geomagic) that is used to measure changes and deviations between the scans. The data collected will provide valuable insights into the long-term performance and stability of the different materials used in the full-arch restorations, thereby contributing to the understanding of their clinical efficacy in implant-supported prosthetics.

ELIGIBILITY:
Inclusion Criteria:

* non-smokers
* patients with adequate bone height and width
* patients with good oral hygiene and healthy gingiva

Exclusion Criteria:

* smokers
* patients with inadequate bone height and width
* non-compliant patients
* patients with systemic diseases that will affect bone remodelling

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2025-08-08 (Estimated); Study Completion 2025-08-08 (Estimated)

PRIMARY OUTCOMES:
bone height changes around the implants | 12 months
  bone height changes around the implants will be assessed using CBCT. this will be acquired at the time of insertion, after 6 months and after 12 months. bone height changes will be measured at the buccal, mesial, distal and lingual surfaces around each implant.

SECONDARY OUTCOMES:
occlusal surface wear analysis | 12 months
  occlusal surface wear analysis will be performed by taking intraoral scans and saving the scan (STL) files to be imported into a specific software that is used to compare and measure the deviations between the reference file and the new files. the scans will be taken at the time of framework insertion, after 6 months and after 12 months post-insertion.

CONTACTS AND LOCATIONS:
Locations (1):
- Misr University for Science and Technology, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all IPD collected throughout the trial, only IPD used in the results publication
Supporting Information: Study Protocol, CSR
Time Frame: starting 6 months after publication
Access Criteria: practitioners interested in the same field of research
URL: https://clinicaltrials.gov